CLINICAL TRIAL: NCT02483299
Title: Liraglutide as Add on Therapy on Metformin in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Andrej Janez, professor, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIRA COMBI
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: PCOS; Obesity
Keywords: response to therapy
MeSH Terms: conditions — Obesity | interventions — Metformin; Liraglutide; Solutions; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- metformin (Active Comparator): In the metformin group metformin was initiated at a dose of 500 mg once per day and increased by 500 mg every 3 days up to 1000 mg BID per os.
  Interventions: Drug: Metformin
- combined (Active Comparator): In the metformin and liraglutide group metformin was initiated at a dose of 500 mg once per day and increased by 500 mg every 3 days up to 1000 mg BID per os. At the same time liraglutide was initiated at a dose of 0.6 mg injected sc once per day and increased to 1.2 mg/day after 1 week.
  Interventions: Drug: Glucophage tablets and Victoza

INTERVENTIONS:
Drug: Metformin
  Other Names: Glucophage tablets
  Arms: metformin
Drug: Glucophage tablets and Victoza
  Other Names: Glucophage tablets and Victoza 6 mg/ml solution for injection in pre-filled pen
  Arms: combined

SUMMARY:
The purpose of this study was to determine whether combined treatment with liraglutide and metformin is more effective than metformin as monotherapy in the treatment of obese women with polycystic ovary syndrome (PCOS). We anticipated greater changes in body weight in patients on combined treatment than in those on monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old to menopause
* polycystic ovary syndrome (NICHD criteria)
* BMI of 30 kg/m² or higher

Exclusion Criteria:

* type 1 or type 2 diabetes mellitus
* history of carcinoma
* Cushing's syndrome or congenital (non-classic) adrenal hyperplasia
* personal or family history of MEN 2
* significant cardiovascular, kidney or hepatic disease
* the use of medications known or suspected to affect reproductive or metabolic functions
* the use of statins, within 90 days prior to study entry

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in body weight | up to 12 weeks of clinical trial
The number of good responders to combined treatment regarding body weight | up to 12 weeks of clinical trial

SECONDARY OUTCOMES:
Change in body mass index (BMI). | up to 12 weeks of clinical trial
  Patient's BMI was defined as the patient's body mass in kilograms divided by the square of their height in meters.
Change in waist circumference | up to 12 weeks of clinical trial
  waist circumference was measured in centimeters.

OTHER OUTCOMES:
Change in fasting concentrations of glucose | up to 12 weeks of clinical trial
  Patient's blood was drawn between 8 and 9 a.m. Concentrations of fasting glucose was measured in mmol/L.
Change in fasting concentration of insulin | up to 12 weeks of clinical trial
  Patient's blood was drawn between 8 and 9 a.m. Fasting concentrations of insulin was measured in mU/L.
Change in blood concentrations of LH (luteinizing hormone) | up to 12 weeks of clinical trial
  Patient's blood was drawn between 8 and 9 a.m. Concentration of LH was measured in U/L.
Change in blood concentrations of FSH (follicle-stimulating hormone) | up to 12 weeks of clinical trial
  Patient's blood was drawn between 8 and 9 a.m. Blood concentrations of FSH was measured in U/L.
Change in blood concentration of testosterone | up to 12 weeks of clinical trial
  Patient's blood was drawn between 8 and 9 a.m. Blood concentration was measured in nmol/L.
Change in blood concentration in androstenedione | up to 12 weeks of clinical trial
  Patient's blood was drawn between 8 and 9 a.m. Blood concentrations of androstenedione was measured in nmol/L.
Change in blood concentrations of SHBG (sex hormone-binding globulin) | up to 12 weeks of clinical trial
  Patient's blood was drawn between 8 and 9 a.m. Blood concentrations of SHBG was measured in nmol/L.
Change in blood concentration of DHEAS (dehydroepiandrosterone sulfate) | up to 12 weeks of clinical trial
  Patient's blood was drawn between 8 and 9 a.m. Blood concentrations of DHEAS was measured in micromol/L.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia